CLINICAL TRIAL: NCT04682236
Title: Study of the Evolution Profile of the Renal Doppler in the Perioperative Hepathic Transplantation - Interest in Predicting the Occurence of Acute Postoperative Renal Faillure
Brief Title: Study of the Evolution Profile of the Renal Doppler in the Perioperative Hepathic Transplantation
Acronym: DOP-RENAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8059
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Acute Renal Failure
Keywords: Acute Renal Failure; Chronic renal failure; Liver transplant; Renal vascular profiles; Intraoperative hemodynamic instability; Acute tubular necrosis; Renal doppler
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Kidney Cortex Necrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplantation is associated with a modification of the perfusion pressures of the abdominal organs (preoperative portal hypertension in connection with liver pathology, and normalization of the perfusion pressures during surgery). This abrupt change in the infusion regime is probably responsible for an alteration in renal function in some patients, and the identification of renal vascular profiles using Doppler could point to pathological profiles, which should be diagnosed early.

ELIGIBILITY:
Inclusion Criteria:

* Patient of full age (≥18 years)
* Patient operated on at the HUS for a liver transplant, between July 1, 2019 and June 30, 2020.
* Patients having undergone an evaluation of hepatic and renal vascular profiles perioperatively.
* Patients hospitalized in the surgical intensive care unit after hepatic transplant surgery.
* Patient not having expressed, after information, the reuse of his data for the purposes of this research

Exclusion Criteria:

* Patient who expressed his opposition to participating in the study
* Patient with suspected obstructive acute renal failure
* Stenosis of renal arteries known at the time
* End-stage renal disease on dialysis
* Impossibility of giving the subject informed information (difficulties in understanding the subject, etc.)
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient operated on at the HUS for a liver transplant, between July 1, 2019 and June 30, 2020
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-05-25 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of the development profiles of renal dopplers in perioperative liver transplantation | Files analysed retrospectily from July 1st, 2019 to June 30, 2020 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Julien POTTECHER, MD, PhD, Study Director — Strasbourg University Hospitals - Anesthesia-intensive care unit
Locations (1):
- Strasbourg University Hospitals - Anesthesia-intensive care unit, Strasbourg, France